CLINICAL TRIAL: NCT06027684
Title: Intensive Care Decision-making, Survival and Dying Well: How do the Experiences of Intensive Care Patients and Their End-of-life Wishes Affect Their Willingness to Accept Intensive Care Treatment at Different Chances of Survival?
Brief Title: Intensive Care Decision-making, Survival and Dying Well
Status: Recruiting | Type: Observational
Sponsor: University of Manchester (Other)
Collaborators: The Royal College of Anaesthetists (Other)
Responsible Party: Principal Investigator, Thomas Donaldson, PhD Student, University of Manchester
Other Study IDs: NHS002026; 317639 (Other: IRAS ID)
Record Dates: First submitted 2023-08-09; First posted 2023-09-07 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to investigate how the experiences of intensive care patients and their end-of-life wishes affect their willingness to accept intensive care treatment at different chances of survival.

The main questions it aims to answer are:

* What can ICU survivors' experiences of ICU treatment tell us about what it would be like to die whilst receiving ICU treatment?
* How do ICU survivors' reflections about what it might be like to die on ICU relate to their own preferences for their end-of-life care?
* What chance of survival would make ICU survivors willing to go through ICU treatment again, in light of the fact that the alternative chance is dying whilst experiencing ICU treatment?
* How does the possibility of reduction in health-related quality of life and functional decline as a result of critical illness impact ICU survivors' willingness to accept ICU treatment again?

Participating in this study will involve filling out a questionnaire and then taking part in an interview. Participants will be recruited through ICU review clinics and ICU steps groups. The study will last for two years and will be conducted at locations convenient to the participants or via zoom.

DETAILED DESCRIPTION:
The ageing population of many countries has led to more elderly and increasingly co-morbid patients accessing healthcare services, and intensive care is no exception. This creates an increasing demand for intensive care treatment for patients with a low chance of surviving their critical illness, even with intensive care treatment.

A sedated intensive care patient receiving mechanical ventilation may have the appearance of being unconscious, but follow-up studies with survivors show that many patients have memories of their experiences, which have been described as frightening and chaotic, leading to feelings of instability, vulnerability and fear. Studies have reported recall of pain, disturbing dreams, procedures, thirst, noise, difficulty communicating, difficulty swallowing, awareness of invasive tubes, panic/fear, helplessness, lack of control, feeling tense and patients thinking they were dying. In one study, 67% of patients had recollections of stressful experiences whilst receiving intensive care treatment and 66-92% of these experiences were rated as moderately to extremely distressing. It must be assumed that all intensive care patients (survivors and non-survivors) have similar experiences of their treatment. Therefore, the negative experiences described by survivors must be assumed to be shared by patients who die whilst receiving such treatment. Consequently, dying whilst receiving intensive care treatment is likely to be a significantly distressing experience.

Intensive care treatment may not be beneficial for patients with a low chance of surviving critical illness if the treatment has a high chance of exposing them to a negative dying experience. For intensive care treatment to be ethically justifiable it should offer patients a reasonable chance of survival to justify the burdens inherent in the treatment, and the risks of a negative dying experience. Therefore, a key question in the provision of intensive care treatment is at what chance of survival is this treatment ethically justifiable? An adequate answer to this question will require consideration of both the quantitative benefits of the treatment, such as survival, and the qualitative harms, including suffering and the risk of exposure to a negative dying experience.

Even though dying whilst receiving intensive care treatment is likely to be a negative dying experience, it is not possible to ask patients who did not survive their critical illness about their dying experience or whether they retrospectively agree with the decision to provide them with intensive care treatment. However, all intensive care patients (survivors and non-survivors) have experiences of what it is like to receive intensive care treatment. All ICU patients can be considered a population whose experiences can be represented by the survivors of ICU. Therefore, the experiences described by survivors can provide a window into the experience of patients who die whilst receiving such treatment.

Research to establish the harm-to-benefit ratio that most people would be willing to accept with regards to intensive care treatment is, therefore, of great importance to guide ethical decision-making regarding the provision of intensive care treatment. Of particular importance will be elderly and co-morbid patients' evaluations of their negative intensive care experiences, as these patients are likely to be the ones with the lowest chance of surviving a critical illness. This information could be used to guide intensive care decision-making and to better inform patients of the harms of intensive care treatment. Such research could provide guidance regarding what chance of survival makes the suffering involved in intensive care treatment, acceptable to patients and ensure that intensive care treatment is not routinely offered to patients with a very low chance of surviving their critical illness, for whom the benefit does not outweigh the cost.

ELIGIBILITY:
Inclusion Criteria:

* The principle inclusion criteria are being 18 years or older and having previously been a patient on an intensive care/critical care unit in the past.
* Being willing to talk about experiences of intensive care treatment, end-of-life wishes, and the context (chances of survival/functional decline) which would make intensive care treatments acceptable and being willing to either meet in person or have access to a computer, tablet or mobile phone with video and a stable internet connection (for a Zoom conversation) are also inclusion criteria.

Exclusion Criteria:

* The exclusion criteria are being under the age of 18, having had a planned admission to an intensive care/critical care unit (e.g. after an elective operation), being unable to consent to participate in the research and having a significant language barrier (as there is no available funding to pay for translation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (over the age of 18) participants who have experience as a patient on an intensive care/critical care unit will be recruited in this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The chance of survival that would make participants willing to go through critical care treatment again. | 2 years
  The mixed methods approach will involve triangulation of qualitative and questionnaire data about participants' experiences of intensive care treatment, end-of-life wishes, and the chance of survival that would make them willing to go through critical care treatment again.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Donaldson, MB/BChir, Principal Investigator — University of Manchester
Locations (1):
- University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
At the end of the project, the investigators will deposit a fully anonymised dataset [e.g., including de-identified interview transcripts] in an open data repository where it will be permanently stored. The investigators will use Figshare at the University of Manchester Library. Researchers at other institutions and others can access the anonymised data directly from the repository and use it for further research or to check the analysis and results. Participants are informed of this in the participant information sheet and will be asked to consent to this on the consent form.
Time Frame: At the end of the study.

DOCUMENTS (2):
  • Study Protocol (2023-04-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT06027684/Prot_000.pdf
  • Informed Consent Form (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT06027684/ICF_001.pdf